CLINICAL TRIAL: NCT01571063
Title: Treatment of Non-alcoholic Steatohepatitis (NASH) Patients With Vitamin D
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SASL 34
Record Dates: First submitted 2012-03-28; First posted 2012-04-04 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Non-alcoholic Steatohepatitis (NASH)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Vitamin D3 (Experimental)
  Interventions: Drug: Vitamin D3; Drug: Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: Vitamin D3; Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D3 — Vitamin D3, 2.100 IU/d p.o.
Drug: Placebo — Placebo Tbl. p.o.

SUMMARY:
Test the efficacy of vitamin D to improve non-alcoholic steatohepatitis with regard to biochemical and histological parameters.

* Trial with medicinal product

ELIGIBILITY:
Inclusion criteria:

* Patients with 25-OH vitamin D insufficiency
* Elevated alanine aminotransferase level
* Diagnosis of definite or possible steatohepatitis (NASH)

Exclusion criteria:

* Cirrhosis, present liver disease other than NASH
* Serious diseases limiting life expectancy,
* Breast-feeding or pregnant women
* Unhealthy alcohol consumption
* Drug abuse or substitution therapy
* Use of vitamin preparations within the previous 6 months and during the study
* Weight loss >5% within 12 months before study entry
* Newly diagnosed Diabetes mellitus requiring medical treatment within 12 months before study entry
* Use of anti-obesity drugs
* Previous or current hypercalcemia
* Chronic renal disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in serum alanine aminotransferase levels at week 48 | Measurement at week 0 and week 48

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Geier, Prof. MD, Study Director — University Hospital Zurich, Division of Hepatology; Beat Muellhaupt, Professor, MD, Principal Investigator — University Hospital Zurich, Division of Gastroenterology and Hepatology
Locations (2):
- Switzerland (2):
  - University Hospital Zurich, Gastroenterology and Hepatology, Zurich, Canton of Zurich
  - Kantonsspital St. Gallen, Sankt Gallen